CLINICAL TRIAL: NCT03559491
Title: Evaluation of the Effectiveness of Treatment With Dexamethasone Intravitreal Implant in Cystoid Macular Edema Secondary to Retinal Vein Occlusion
Brief Title: Dexamethasone Intravitreal Implant in Retinal Vein Occlusion
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Simone Donati, Study Investigator, Università degli Studi dell'Insubria
Other Study IDs: 2018oculistica
Record Dates: First submitted 2018-06-05; First posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-06

CONDITIONS: Macular Edema, Cystoid
Keywords: steroid; retinal vein occlusion; macular edema
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Intravitreal Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Macular Edema Patients: Patients affected by cystoid macular edema (CME) due to retinal vein occlusion of recent onset (less than three months) will be enrolled.
  Interventions: Drug: Intravitreal injection

INTERVENTIONS:
Drug: Intravitreal injection — Long term release steroid injection

SUMMARY:
Purpose: To evaluate retinal functional improvement by means of visual acuity and retinal sensibility examination after intravitreal dexamethasone implant in patients affected by cystoid macular edema secondary to retinal vein occlusion.

DETAILED DESCRIPTION:
Cystoid macular edema represents the most important cause of visual impairment after retinal vein occlusion. The etiological factors of this complication are under investigation, from inflammatory cytokines to the breakdown of vascular barrier with increased permeability and diffusion of angiogenic factors. Clinical research developed different drugs and therapeutic strategies to treat and control macular edema, to evaluate the correct timetable and to reach long-term clinical significative results. At now, different experiences have been published with available drugs, from steroids to anti Vascular Endothelial Growth Factor. A debate still remains about the correct approach, the correct combination of drugs (if necessary) and the correct evaluation of drug effectiveness.

In our study, we will evaluate extensive functional recovery and its relation to macular thickness after steroid injection. Considering that visual acuity reflects only foveal function, it may not be sufficient to evaluate the overall function on the macular area. We introduce microperimetry study as a valuable and reproducible tool to create a functional mapping of the entire macula.

ELIGIBILITY:
Inclusion criteria were: age older than 18 years; CME secondary to retinal vein occlusion, disease duration inferior to 12 weeks; best-corrected visual acuity (BCVA) between 20/200 and 20/25 (Snellen equivalent) in the study eye at baseline examination, central retinal thickness (CRT) superior to 300 mm, as measured by optical coherence tomography at baseline examination.

The exclusion criteria were any ocular surgery in the study eye in the past 6 months; diabetes mellitus with signs of diabetic retinopathy; previous laser photocoagulation; previous intravitreal injection of corticosteroids or anti-vascular endothelial growth factor; a history of ocular inflammation; marked retinal ischemia or retinal hemorrhages (in particular in macular region involving the fovea); any other ocular condition such as anterior ischemic neuropathy, amblyopia or significant media opacities; significant alteration on epiretinal surface such as epiretinal membrane or vitreomacular traction; uncontrolled or advanced glaucoma; any uncontrolled systemic disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by cystoid macular edema (CME) due to retinal vein occlusion of recent onset (less than three months) were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 6 months
  evaluation of visual acuity
retinal sensibility | 6 months
  microperimetry evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Simone Donati, MD, Principal Investigator — Università dell'Insubria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Querques G, Lattanzio R, Querques L, Triolo G, Cascavilla ML, Cavallero E, Del Turco C, Casalino G, Bandello F. Impact of intravitreal dexamethasone implant (Ozurdex) on macular morphology and function. Retina. 2014 Feb;34(2):330-41. doi: 10.1097/IAE.0b013e31829f7495. PMID 23945638
- [Result] Garweg JG, Zandi S. Impact of treatment on long-term visual function in retinal vein occlusion-response to the comment on: retinal vein occlusion and the use of a dexamethasone intravitreal implant (Ozurdex(R)) in its treatment. Graefes Arch Clin Exp Ophthalmol. 2016 Dec;254(12):2479-2480. doi: 10.1007/s00417-016-3459-y. Epub 2016 Sep 7. No abstract available. PMID 27604764
- [Derived] Donati S, Gandolfi C, Caprani SM, Cattaneo J, Premoli L, Azzolini C. Evaluation of the Effectiveness of Treatment with Dexamethasone Intravitreal Implant in Cystoid Macular Edema Secondary to Retinal Vein Occlusion. Biomed Res Int. 2018 Aug 2;2018:3095961. doi: 10.1155/2018/3095961. eCollection 2018. PMID 30175123